CLINICAL TRIAL: NCT02601599
Title: Medical Student INtervention to Promote Effective Nicotine Dependence and Tobacco HEalthcare: GrAduate Entry Programme (MIND-THE-GAP) Feasibility Randomised Trial
Brief Title: Medical Student INtervention to Promote Effective Nicotine Dependence and Tobacco HEalthcare
Acronym: MIND-THE-GAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Health Service Executive, Ireland (Other); University of Memphis (Other); Connolly Hospital Blanchardstown (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC1126
Record Dates: First submitted 2015-11-03; First posted 2015-11-10 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2016-04

CONDITIONS: Smoking
Keywords: Smoking Cessation; Tobacco Use Cessation; Motivational Interviewing; Students, Medical; Randomized Controlled Trial
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Cessation | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Motivational interviewing The medical student will deliver a 15 minute consultation with the patient. The goals of this consultation will be to enhance the patient's motivation and self-efficacy regarding quitting, educate the patient about effective behavioral and pharmacological cessation strategies, and collaboratively elicit a plan to stay quit after discharge. Patients will be offered the opportunity to receive a consultation from the attending physician to determine eligibility for pharmacotherapy. Patients who elect to receive this consult with have a coloured sticker placed by the medical student on the medical chart requesting a consultation.
  Interventions: Behavioral: Motivational interviewing
- Usual care (No Intervention): This group will not receive student contact, but may be counselled by the smoking cessation officer or other Connolly staff as per normal procedures.

INTERVENTIONS:
Behavioral: Motivational interviewing — The medical student will deliver a brief (approximately 15 minute) consultation with the patient that is based on principles of social cognitive theory and motivational interviewing. The goals of this consultation will be to enhance the patient's motivation and self-efficacy regarding quitting, and collaboratively elicit a plan to stay quit after discharge. Patients will be offered the opportunity to receive a consultation from the attending physician to determine eligibility for pharmacotherapy (via a chart sticker).
  Each student will counsel 1-3 smokers each over the 8-month academic period, with student training and intervention staggered over this time. Students will also re-contact the smoker at 1-week post-discharge via telephone or personal follow-up, to provide further support.
  Arms: Intervention

SUMMARY:
Background: Smoking counselling during hospitalisation with post-discharge follow-up increases quitting. However, provision of cessation care for hospitalised patients is suboptimal. Students are potentially an untapped resource for providing cessation advice, but no studies have investigated this.

Aim: To determine if medical students can encourage motivation to stop smoking (MTSS; primary outcome) in hospitalised smokers .

Design: 2-arm RCT Setting: RCSI (www.rcsi.ie) and Connolly Hospital (www.hse.ie/eng/services/list/3/hospitals/Connolly/).

Participants: Inpatient smokers. Intervention and procedures: 60 graduate medical students will receive standardised motivational interviewing training in the provision of cessation advice. Each student will be randomly assigned to counsel ~1-3 smokers each, including an individual in-hospital, face-to-face session and post-discharge phone counselling. Training and implementation will cover Sept-2015-May-2016. Smokers will be randomised to 'usual care' (n~90), or intervention (n~90, student-delivered motivational interviewing). A researcher will enable recruitment and follow-up, and conduct a qualitative evaluation of programme participants.

ELIGIBILITY:
Inclusion Criteria:

* All identified inpatient smokers at Connolly Hospital.

Exclusion Criteria:

* Advised by ward manager that patient is too unwell or cognitively impaired, or otherwise unsuitable;
* Death during hospitalisation;
* Receiving palliative care;
* Under 18 years of age;
* To be transferred to another hospital;
* Not English speaking;
* Refusal to participate;
* Inpatient in psychiatric ward

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Motivation to Stop Smoking Scale (MTSS) | Repeated measures: MTSS scores at baseline, 1-week, 3- and 6-month follow-up.
  Repeated measures: MTSS scores at baseline, 1-week, 3- and 6-month follow-up.
Change in motivation to quit | Repeated measures: single item scores at baseline, 1-week, 3- and 6-month follow-up.
  If, on a scale of 1 to 10, 1 is not at all motivated to give up smoking and 10 is 100% motivated to give up, what number would you give yourself at the moment?

SECONDARY OUTCOMES:
Proportion of patients who receive a prescription for a cessation medication at the time of discharge | By discharge, an average of 5-10 days post-admission
  The proportion of patients who receive a prescription for a cessation medication at the time of discharge, assessed via medical chart audit;
proportion of patients who report any use of a prescribed or over-the-counter cessation medication | at 3- and 6-months discharge
  the proportion of patients who report any use of a prescribed or over-the-counter cessation medication, of an approved cessation pharmacotherapy, including nicotine patch, gum, lozenge, inhaler, mouth spray, Champix, or Zyban at 1- and 6-months discharge
proportion of attending physicians who prescribe cessation medication during the hospitalisation | During hospitalisation (baseline)
  the proportion of attending physicians who prescribe cessation medication during the hospitalisation (to be obtained by medical chart audit);
7-day point prevalent abstinence rates | 3- and 6-months
  7-day point prevalent abstinence rates assessed at both 3- and 6-months by self-report

OTHER OUTCOMES:
Perceived student efficacy | 3- and 6-months
  Single items survey: How helpful was the support that you received from the medical student?" [not at all, a little bit, somewhat, quite a bit, or very much]?"
Perceived student knowledge | 3- and 6-months
  Single item survey: How knowledgeable was the medical student about quitting smoking? [not at all, a little bit, somewhat, quite a bit, or very much]
Quit attempts | 3- and 6-months
  Three questionnaire items:
  1. In the past one/six months, have you quit smoking? Yes/No
  2. If no, in the past one/six months have you attempted to quit smoking? Yes/No
  3. If yes, how many times have you tried to quit in the past three/six months? ______
Professional advice | 3- and 6 months
  One questionnaire item: In the past 3/6 months since your hospital admission, did a doctor or health professional discuss ways of giving up smoking with you?

CONTACTS AND LOCATIONS:
Overall Officials: Seamus Sreenan, Study Director — RCSI and Connolly Hospital; Liam Cormican, Study Director — RCSI and Connolly Hospital; Ken Ward, Study Director — University of Memphis; Lisa Mellon, PhD, Study Director — RCSI; Ronan Conroy, Study Director — RCSI; Anne Hickey, PhD, Study Director — RCSI; Sinead Stynes, Study Director — Connolly Hospital; Frank Doyle, PhD, Principal Investigator — RCSI; GEP IC1, Study Director — RCSI students
Locations (1):
- Connolly Hospital Blanchardstown, Dublin, Ireland

REFERENCES:
- [Background] 1. Hickey P, Evans DS: Smoking in Ireland 2014: Synopsis of key patterns. In. HSE National Tobacco Control Office, Health and Wellbeing Division: Health Services Executive; 2015.
- [Background] 2. Department of Health: Tobacco Free Ireland: Report of the Tobacco Policy Review Group. In. Dublin: Department of Health; 2013.
- [Background] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. The Health Consequences of Smoking-50 Years of Progress: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2014. Available from http://www.ncbi.nlm.nih.gov/books/NBK179276/ PMID 24455788
- [Background] 4. Bridgehead International: EQUIPP: Europe Quitting: Progress and Pathways. In. London; 2011.
- [Background] Carson KV, Verbiest ME, Crone MR, Brinn MP, Esterman AJ, Assendelft WJ, Smith BJ. Training health professionals in smoking cessation. Cochrane Database Syst Rev. 2012 May 16;2012(5):CD000214. doi: 10.1002/14651858.CD000214.pub2. PMID 22592671
- [Background] Rigotti NA, Clair C, Munafo MR, Stead LF. Interventions for smoking cessation in hospitalised patients. Cochrane Database Syst Rev. 2012 May 16;5(5):CD001837. doi: 10.1002/14651858.CD001837.pub3. PMID 22592676
- [Background] Rigotti NA, Regan S, Levy DE, Japuntich S, Chang Y, Park ER, Viana JC, Kelley JH, Reyen M, Singer DE. Sustained care intervention and postdischarge smoking cessation among hospitalized adults: a randomized clinical trial. JAMA. 2014 Aug 20;312(7):719-28. doi: 10.1001/jama.2014.9237. PMID 25138333
- [Background] O'Donovan G. Smoking prevalence among qualified nurses in the Republic of Ireland and their role in smoking cessation. Int Nurs Rev. 2009 Jun;56(2):230-6. doi: 10.1111/j.1466-7657.2008.00700.x. PMID 19646173
- [Background] Bartels C, Abuhaliga AR, McGee H, Morgan K, McElvaney NG, Doyle F. A survey of the prevalence of smoking and smoking cessation advice received by inpatients in a large teaching hospital in Ireland. Ir J Med Sci. 2012 Sep;181(3):445-9. doi: 10.1007/s11845-011-0792-3. Epub 2012 Jan 6. PMID 22223193
- [Background] Fitzpatrick P, Gilroy I, Doherty K, Corradino D, Daly L, Clarke A, Kelleher CC. Implementation of a campus-wide Irish hospital smoking ban in 2009: prevalence and attitudinal trends among staff and patients in lead up. Health Promot Int. 2009 Sep;24(3):211-22. doi: 10.1093/heapro/dap020. Epub 2009 Jun 16. PMID 19531558
- [Background] 11. Ohakim A, Mellon L, Jafar B, O'Byrne C, McElvaney NG, Cormican L, McDonnell R, Doyle F: Smoking, attitudes to smoking and provision of smoking cessation advice in two teaching hospitals in Ireland: do smoke-free policies matter? Health Psychology and Behavioral Medicine: An Open Access Journal 2015, 3(1):142-153.
- [Background] 12. Mellon L, McElvaney NG, Cormican L, Hickey A, Conroy R, Ekpotu L, Oghenejobo O, Atteih S, McDonnell R, Doyle F: Determining rates of smoking cessation advice delivered during hospitalisation and smoking cessation rates 3-months post discharge: a two-hospital survey. manuscript submitted for publication.
- [Background] Raupach T, Shahab L, Baetzing S, Hoffmann B, Hasenfuss G, West R, Andreas S. Medical students lack basic knowledge about smoking: findings from two European medical schools. Nicotine Tob Res. 2009 Jan;11(1):92-8. doi: 10.1093/ntr/ntn007. Epub 2009 Jan 27. PMID 19246446
- [Background] Raupach T, Merker J, Hasenfuss G, Andreas S, Pipe A. Knowledge gaps about smoking cessation in hospitalized patients and their doctors. Eur J Cardiovasc Prev Rehabil. 2011 Apr;18(2):334-41. doi: 10.1177/1741826710389370. Epub 2011 Feb 11. PMID 21450679
- [Background] Kotz D, Brown J, West R. Predictive validity of the Motivation To Stop Scale (MTSS): a single-item measure of motivation to stop smoking. Drug Alcohol Depend. 2013 Feb 1;128(1-2):15-9. doi: 10.1016/j.drugalcdep.2012.07.012. Epub 2012 Sep 1. PMID 22943961
- [Background] West R, Hajek P, Stead L, Stapleton J. Outcome criteria in smoking cessation trials: proposal for a common standard. Addiction. 2005 Mar;100(3):299-303. doi: 10.1111/j.1360-0443.2004.00995.x. PMID 15733243
- [Background] Arora NK, Gustafson DH. Perceived helpfulness of physicians' communication behavior and breast cancer patients' level of trust over time. J Gen Intern Med. 2009 Feb;24(2):252-5. doi: 10.1007/s11606-008-0880-x. Epub 2008 Dec 17. PMID 19089501
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] 19. Freidman LM, Furberg CD, DeMets DL: Fundamentals of Clinical Trials, 4th Edition edn. New York: Springer; 2010.
- [Derived] Kumar A, Ward KD, Mellon L, Gunning M, Stynes S, Hickey A, Conroy R, MacSweeney S, Horan D; Graduate Entry Programme 2014-18 Class; Cormican L, Sreenan S, Doyle F. Medical student INtervention to promote effective nicotine dependence and tobacco HEalthcare (MIND-THE-GAP): single-centre feasibility randomised trial results. BMC Med Educ. 2017 Dec 11;17(1):249. doi: 10.1186/s12909-017-1069-y. PMID 29233157